CLINICAL TRIAL: NCT06044597
Title: Post-market Prospective, Multicenter, Randomized and Single-blinded Clinical Investigation to Evaluate Whether Cardiac Re-Synchronization Therapy (CRT) Using Automatic Continuous Atrioventricular (AV) Delay Optimization is Superior to CRT With Conventional Biventricular Stimulation (BiV). (CRUSTY + Trial)
Brief Title: Post-market Prospective, Multicenter, Randomized and Single-blinded Clinical Investigation to Evaluate Whether Cardiac Re-Synchronization Therapy (CRT) Using Automatic Continuous Atrioventricular (AV) Delay Optimization is Superior to CRT With Conventional Biventricular Stimulation (BiV).
Acronym: CRUSTY +
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Antonio Rapacciuolo (Other)
Responsible Party: Sponsor-Investigator, Antonio Rapacciuolo, Principal Investigator, Federico II University
Organization: Federico II University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DE-66-22
Record Dates: First submitted 2023-08-07; First posted 2023-09-21 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2023-09

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Intervention Model Description: Randomized study with 2 groups: control group (Traditional biventricular stimulation), study group (biventricular stimulation + SyncAV feature)
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SyncAV plus group (Experimental): Patients implanted with a CRT-D programmed with SyncAV plus function ON.
  Interventions: Device: SyncAV function on
- Biv Trad (No Intervention): Patients implanted with a CRT-D programmed with fixed AV delay.

INTERVENTIONS:
Device: SyncAV function on — CRT-D with SyncAV plus activated
  Arms: SyncAV plus group

SUMMARY:
The goal of this randomized, multicenter prospective study is to demonstrate that the activation of biventricular pacing with fusion and AV optimization feature will increase the rate of CRT responders in terms of LV reverse remodeling, compared with conventional biventricular pacing.

DETAILED DESCRIPTION:
Treatment of HFrEF with CRT. CRT is an established guideline-recommended treatment for patients who are refractory to optimized pharmacologic therapy, and have reduced ejection fraction and increased QRS duration. It works by restoring atrioventricular, inter- and intra-ventricular synchrony and in so doing, it has been shown to improve symptoms, LV systolic function and survival. Nevertheless, a significant proportion of patients (30-45%) do not benefit after CRT and are considered non-respondent. Non-response to CRT is multifactorial (poor substrate to resynchronize, difficulty in the implant, age, gender, aetiology, and/or comorbidities). Recently, other negative determinants have been identified as cause of non-responding to CRT such as the lack of fusion of ventricular contraction with the intrinsic right ventricular conduction and non-optimal AV delay programming which, in turn, is related to the duration of PR interval. Another possible reason for non-responding to CRT is a non-optimal LV pacing site.

The CRUSTY PLUS trial is aimed to establish the relevance for the success of CRT of these three factors: lack of fusion, non-optimized A-V conduction, and LV pacing site by comparing the response to CRT with a standard BIV device with fixed out-of-the-box A-V delay with that to a BIV device (Sync A-V plus) endowed with an algorithm which is continuously measuring the patients' A-V conduction and is able to adjust the stimulation parameters according to the measured PR interval, achieving a more dynamic A-V interval and allowing a perfect fusion of ventricular contraction. The algorithm is also able to optimize LV intraventricular synchrony. Sync A-V plus is endowed with a quadripolar multipoint pacing (MPP) CRT-D system allowing pacing of the LV with 2 vectors. This methodology allows a simultaneous earlier and wider excitation of ventricular tissue resulting in better synchronization and better cardiac output.

ELIGIBILITY:
Inclusion Criteria:

* More than 18 years of age;
* Have signed the Informed Consent form.
* have been implanted with an Abbott CRT-D with the Sync-AV dynamic function under the current Class I or Class IIa ESC indications (2021 guidelines) for CRT implantation (including upgrades from single or dual chamber pacemakers or ICDs);
* Have to be in sinus rhythm at the Baseline visit and with Left Branch Block (LBBB) (2021 ESC/REVERSE):
* LVEF needs to be <35% while under optimal medical treatment
* to be willing to meet all study requirements and have the ability to do participate to this study.

Exclusion Criteria:

Inclusion / Exclusion criteria: Inclusion criteria: To participate in this clinical study, patients must meet ALL of the following inclusion criteria:

* More than 18 years of age;
* Have signed the Informed Consent form.
* And have been implanted with an Abbott CRT-D with the Sync-AV dynamic function under the current Class I or Class IIa ESC indications (2021 guidelines) for CRT implantation (including upgrades from single or dual chamber pacemakers or ICDs);
* Have to be in sinus rhythm at the Baseline visit and with Left Branch Block (LBBB) (2021 ESC/REVERSE):
* LVEF needs to be <35% while under optimal medical treatment
* In addition, patients need to be willing to meet all study requirements and have the ability to do participate to this study.

Exclusion criteria: Patients who meet any of the following exclusion criteria are NOT eligible to participate in the clinical study:

* Having suffered a myocardial infarction or unstable angina in the 40 days prior to inclusion.
* Having undergone coronary revascularization (PTCA, Stent or CABG) in the 4 weeks prior to inclusion.
* Having suffered a Cerebrovascular Accident (CVA) or a Transient Ischemic Accident (TIA) in the 3 months prior to inclusion.
* NYHA Class IV.
* Having received a heart transplant or being waiting to receive it (status I classification);
* Suffering from primary valve disease requiring surgical intervention.
* Having long-lasting or permanent atrial fibrillation
* Showing inadequate transthoracic echocardiographic images which will not allow to establish cardiac output and LV volumes.
* Having a life expectancy <12months.
* Being pregnant or planning to become pregnant during the clinical investigation.
* Inability to meet the monitoring schedule.
* Currently participating in any other clinical interventional research.
* Having a permanent high degree AV block

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 722 (Estimated)
Dates: Start 2023-10-01 (Estimated); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-10-30 (Estimated)

PRIMARY OUTCOMES:
Reduction in left ventricular end systolic volume (LVESV) between baseline and 6 months | Month 6
  The primary endpoint is response to CRT defined as > 15% relative reduction in Left Ventricular End Systolic Volume (LVESV) at 6 months after implantation, evaluated by Echocardiography
Reduction in QRS duration after randomization | within 10 days
  The primary endpoint is the reduction of QRS duration compared to the intrinsic QRS.
  Defined as > 13% relative reduction in QRS duration compared with the intrinsic QRS, evaluated by ECG.Defined as > 13% relative reduction in QRS duration compared with the intrinsic QRS, evaluated by ECG.

SECONDARY OUTCOMES:
Percentage of CRT Responders at 12 months after MPP activation programmed after the 6 Months follow-up. | Month 6
  Percentage of non-responders at 6 Months responders at 12 Months with MPP

CONTACTS AND LOCATIONS:
Overall Officials: Jaume Francisco Pascual, Dr, Study Chair — Hospital Vall d'Hebron; Nuria Rivas Gandara, Dr, Study Chair — Hospital Vall d'Hebron; Angelo Auricchio, Prof, Study Chair — Istituto Cardiocentro Ticino